CLINICAL TRIAL: NCT04676685
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Ascending Dose and Single Dose Food Effect Study to Assess the Safety, Tolerability, and Pharmacokinetics of E2730 in Healthy Subjects
Brief Title: A Study to Assess the Safety and Tolerability of E2730 After Multiple Dose and the Food Effect After Single Dose in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: E2730-A001-013
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Healthy Volunteers
Keywords: E2730; Healthy participants; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A, Cohort 1: E2730 20 Milligram (mg) or Placebo (Experimental): Healthy Japanese and non-Japanese participants will receive E2730 20 mg or E2730-matched placebo, capsules, orally, once daily for 18 days under fasted conditions.
  Interventions: Drug: E2730; Drug: E2730-matched placebo
- Part A, Cohort 2: E2730 40 mg or Placebo (Experimental): Healthy Japanese and non-Japanese participants will receive E2730 40 mg or E2730-matched placebo, capsules, orally, once daily for 18 days under fasted conditions.
  Interventions: Drug: E2730; Drug: E2730-matched placebo
- Part A, Cohort 3: E2730 60 mg or Placebo (Experimental): Healthy Japanese and non-Japanese participants will receive E2730 60 mg or E2730-matched placebo, capsules, orally, once daily for 18 days under fasted conditions.
  Interventions: Drug: E2730; Drug: E2730-matched placebo
- Part A, Cohort 4: E2730 80 mg or Placebo (Experimental): Healthy Japanese and non-Japanese participants will receive E2730 80 mg or E2730-matched placebo, capsules, orally, once daily for 18 days under fasted conditions.
  Interventions: Drug: E2730; Drug: E2730-matched placebo
- Part B, E2730 80 mg: Fasted + Fed (Experimental): Participants will receive a single treatment of E2730 (80 mg capsule) in fasted condition on Day 1 treatment period 1 followed by E2730 80 mg capsule in fed condition on Day 1 of treatment period 2. A washout period of at least 21 days will be maintained between the 2 treatments.
  Interventions: Drug: E2730
- Part B, E2730 80 mg: Fed + Fasted (Experimental): Participants will receive a single treatment of E2730 80 mg capsule in fed condition on Day 1 of treatment period 1 followed by E2730 80 mg capsule in fasted condition on Day 1 of treatment period 2. A washout period of at least 21 days will be maintained between the 2 treatments.
  Interventions: Drug: E2730

INTERVENTIONS:
Drug: E2730 — E2730 capsules.
Drug: E2730-matched placebo — E2730-matched placebo capsules.
  Arms: Part A, Cohort 1: E2730 20 Milligram (mg) or Placebo; Part A, Cohort 2: E2730 40 mg or Placebo; Part A, Cohort 3: E2730 60 mg or Placebo; Part A, Cohort 4: E2730 80 mg or Placebo

SUMMARY:
The primary purpose of the study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of E2730 of multiple ascending oral doses in healthy adult participants and to assess the differences in PK, safety, and tolerability of E2730 between healthy Japanese and non-Japanese participants following multiple doses. This study will also determine the effect of food on PK of E2730.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking, healthy male or female, age greater than or equal to (>=) 18 years and <55 years old at the time of informed consent. To be considered non-smokers, Participants must have discontinued smoking for at least 4 weeks before dosing
2. Japanese Participants must have been born in Japan of Japanese parents and Japanese grandparents, must have lived no more than 5 years outside of Japan, and must not have changed their life style or habits, including diet, while living outside of Japan
3. Body mass index (BMI) >=18 and <30 kilograms per meter square (kg/m^2) at Screening

Exclusion Criteria:

1. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [β-hCG] test). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug
2. Females of childbearing potential who:

   * Within 28 days before study entry, did not use a highly effective method of contraception, which includes any of the following:
   * Total abstinence (if it is their preferred and usual lifestyle)
   * An intrauterine device or intrauterine hormone-releasing system (IUS)
   * A contraceptive implant
   * An oral contraceptive (Participant must have been on a stable dose of the same oral contraceptive product for at least 28 days before dosing and must agree to stay on the same dose of the oral contraceptive throughout the study and for 28 days after study drug discontinuation)
   * Have a vasectomized partner with confirmed azoospermia
   * Do not agree to use a highly effective method of contraception throughout the entire study period and for 28 days after study drug discontinuation
3. Males who have not had a successful vasectomy (confirmed azoospermia) if their female partners meet the exclusion criteria above (that is, the female partners are of childbearing potential and are not willing to use a highly effective contraceptive method throughout the study period and for 5 times the half-life of the study drug plus 90 days after study drug discontinuation)
4. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing
5. Evidence of disease that may influence the outcome of the study within 4 weeks before dosing; example, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism
6. Any history of gastrointestinal surgery that may affect PK profiles of E2730, example, hepatectomy, nephrectomy, and digestive organ resection
7. Any clinically abnormal symptom or organ impairment found by medical history, physical examinations, vital signs, ECG finding, or laboratory test results that require medical treatment at Screening
8. A prolonged QT interval of the ECG/Corrected QT interval (QT/QTc) (QTcF greater than [>] 450 milliseconds [ms]) demonstrated by a repeated ECG at Screening or Baseline (based on average of triplicate ECGs). A history of risk factors for torsade de pointes (example, heart failure, hypokalemia, family history of long QT Syndrome) or the use of concomitant medications that prolonged the QT/QTc interval
9. Persistent systolic BP >139 or <90 millimeter of mercury (mmHg) or diastolic BP >89 or <50 mmHg at Screening or Baseline
10. Heart rate <45 beats/minute or >100 beats/minute at Screening or Baseline
11. Any lifetime history of suicidal ideation or any lifetime history of suicidal behavior as indicated by the Columbia-Suicide Severity Rating Scale (C-SSRS) or equivalent scale or via interview with a psychiatrist
12. Any lifetime history of psychiatric disease (including but not limited to depression or other mood disorders, bipolar disorder, psychotic disorders, including schizophrenia, panic attacks, anxiety disorders ). The absence of a history of psychiatric disease should be documented by a checklist in the electronic case report form (eCRF)
13. Any current psychiatric symptoms as indicated by a standard screening tool
14. Any suicidal ideation with intent with or without a plan at Screening or within 6 months of Screening (that is, answering "Yes" to questions 4 or 5 on the Suicidal Ideation section of the C-SSRS)
15. Any lifetime suicidal behavior (per the Suicidal Behavior Section of the C-SSRS)
16. Known history of clinically significant drug allergy at Screening
17. Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening
18. Known to be human immunodeficiency virus (HIV) positive at Screening
19. Active viral hepatitis (A, B, or C) and syphilis as demonstrated by positive serology at Screening
20. History of drug or alcohol dependency or abuse, or those who have a positive drug test at Screening or Baseline
21. Exposure within the last 14 days to an individual with confirmed or probable corona virus disease 2019 (COVID-19) or symptoms within the last 14 days that are on the most recent Centers for Disease Control and Prevention (CDC) list of COVID symptoms or any other reason to consider the participants at potential risk for an acute COVID-19 infection
22. Currently enrolled in another clinical study or used any investigational drug or device within 28 days or 5 half-lives, whichever is longer, preceding informed consent
23. Receipt of blood products within 4 weeks, or donation of blood within 8 weeks, or donation of plasma within 1 week of dosing
24. Any personal or family history of seizures (including febrile seizures) or epilepsy or episode of unexplained loss of consciousness
25. Any history of neurological or other medical conditions which in the opinion of the investigator has the potential to reduce seizure threshold (example, history of head concussion, traumatic brain injury, alcohol abuse, substance abuse, developmental abnormalities in the brain)
26. Any epileptiform discharges on resting EEG (including during hyperventilation and photo-stimulation)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Screening up to Day 32 (approximately 60 days)
  Safety assessments will consist of monitoring and recording all adverse events (AEs); laboratory evaluation for hematology, clinical chemistry, and urinalysis; periodic measurement of vital signs, electrocardiograms (ECGs), electroencephalogram (EEGs), corrected QT (QTc) interval and blood pressure.
Part A, Cmax: Maximum Observed Plasma Concentration for E2730 | Day 1: 0-24 hours; Day 18: 0-336 hours
Part A, Css,min: Minimum Observed Plasma Concentration at Steady State for E2730 | Time Frame: Day 18: 0-24 hours
Part A, tmax: Time at Which the Highest Drug Plasma Concentration Occurs for E2730 | Day 1: 0-24 hours; Day 18: 0-336 hours
Part A, Css,av: Average Steady State Plasma Concentration at Steady State for E2730 | Time Frame: Day 18: 0-24 hours
Part A, AUC(0-24h): Area Under the Plasma Concentration-time Curve From Zero Time to 24 Hours After Dosing for E2730 | Day 1: 0-24 hours; Day 18: 0-24 hours
Part A, t1/2: Terminal Elimination Phase Half-life Following Last day of Dosing for E2730 | Day 18: 0-336 hours
Part A, PTF: Peak-trough Fluctuation for E2730 | Day 18: 0-24 hours
Part A, Rac: Accumulation Ratio for Cmax and AUC for E2730 | Day 1: 0-24 hours; Day 18: 0-24 hours
Part A, CLss/F: Apparent Total Clearance Following Extravascular Administration at Steady State for E2730 | Day 18: 0-336 hours
Part A, Vz/F: Apparent Volume of Distribution at Terminal Phase | Day 18: 0-336 hours
Part B, Cmax: Maximum Observed Plasma Concentration for E2730 | Day 1: 0-288 hours; Day 22: 0-288 hours
Part B, tmax: Time at Which the Highest Drug Plasma Concentration Occurs for E2730 | Day 1: 0-288 hours; Day 22: 0-288 hours
Part B, AUC(0-24h): Area Under the Plasma Concentration-time Curve From Zero Time to 24 Hours After Dosing for E2730 | Day 1: 0-24 hours; Day 22: 0-24 hours
Part B, AUC(0-t): Area Under the Plasma Concentration-time Curve From Zero Time to Time of Last Quantifiable Concentration for E2730 | Day 1: 0-288 hours; Day 22: 0-288 hours
Part B, AUC(0-72h): Area Under the Plasma Concentration-time Curve From Zero Time to 72 Hours After Dosing for E2730 | Day 1: 0-72 hours; Day 22: 0-72 hours
Part B, AUC(0-inf): Area Under the Plasma Concentration-time Curve From Zero Time Extrapolated to Infinite Time for E2730 | Day 1: 0-288 hours; Day 22: 0-288 hours
Part B, t1/2: Terminal Elimination Phase Half-life for E2730 | Day 1: 0-288 hours; Day 22: 0-288 hours
Part A: Geometric Mean Ratio of Cmax Between the Healthy Japanese and non-Japanese Participants for E2730 | Day 1: 0-24 hours; Day 18: 0-336 hours
Part A: Geometric Mean Ratio of AUC(0-24) Between the Healthy Japanese and non-Japanese Participants for E2730 | Day 1: 0-24 hours; Day 18: 0-24 hours
Part B: Geometric Mean Ratio of Cmax Between the Fasted and fed State for E2730 | Day 1: 0-288 hours; Day 22: 0-288 hours
Part B: Geometric Mean Ratio of AUC(0-t) Between the Fasted and fed State for E2730 | Day 1: 0-288 hours; Day 22: 0-288 hours
Part B: Geometric Mean Ratio of AUC(0-72h) Between the Fasted and fed State for E2730 | Day 1: 0-72 hours; Day 22: 0-72 hours
Part B: Geometric Mean Ratio of AUC(0-inf) Between the Fasted and fed State for E2730 | Day 1: 0-288 hours; Day 22: 0-288 hours

SECONDARY OUTCOMES:
Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) | Baseline, Day 32
Change From Baseline in Heart Rate (HR) | Baseline, Day 32
Placebo Corrected Change From Baseline in SBP and DBP | Baseline, Day 32
Placebo Corrected Change From Baseline in HR | Baseline, Day 32
Number of Participants With Categorical Outliers for SBP and DBP | Baseline up to Day 32
Change From Baseline in QT Interval by Fridericia (QTcF) | Baseline, Day 32
Change From Baseline in PR Interval of the ECG (PR), QRS Interval of the ECG (QRS) | Baseline, Day 32
Placebo Corrected Change From Baseline in QTcF, PR and QRS | Baseline, Day 32
Number of Participants With Categorical Outliers for QTcF, HR, PR, and QRS | Baseline, Day 32
Number of Participants With T-wave Morphology Changes | Baseline up to Day 32
  The T-wave morphology categories includes the following: Normal T-wave (Any positive T-wave not meeting any criterion); Flat T-wave (T amplitude less than (<) 1 millimeter [mm] [either positive or negative] including flat isoelectric line); Notched T-wave (+) (Presence of notch(es) of at least 0.05 millivolt [mV] amplitude on ascending or descending arm of the positive T-wave); Biphasic (T-wave that contains a second component with an opposite phase that is at least 0.1 mV deep (both positive/negative and negative/positive and polyphasic T-waves included); Normal T-wave (-) (T amplitude that is negative, without biphasic T-wave or notches); Notched T-wave (-) (Presence of notch(es) of at least 0.05 mV amplitude on descending or ascending arm of the negative T-wave).
Number of Participants With Presence of Abnormal U-wave | Baseline up to Day 32

CONTACTS AND LOCATIONS:
Locations (1):
- Collaborative Neuroscience Research, LLC., Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.